CLINICAL TRIAL: NCT01080404
Title: Obesity, Metabolism and Obstructive Sleep Apnea: Prevalence and the Effect of Bariatric Surgery
Brief Title: A Study of Surgical Weight Loss to Treat Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kuopio University Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other); Turku University Hospital (Other Government); Oulu University Hospital (Other); Vaasa Central Hospital, Vaasa, Finland (Other); Finnish Institute for Health and Welfare (Other Government); Helsingin Uniklinikka (Unknown); Kanta-Häme Central Hospital (Other Government)
Responsible Party: Principal Investigator, Juha Seppa, PhD, MD, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUH5551821
Record Dates: First submitted 2010-03-03; First posted 2010-03-04 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Obstructive Sleep Apnea; Obesity
Keywords: Obstructive sleep apnea; Obesity; Metabolism; Bariatric surgery; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity | interventions — Bariatric Surgery; Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bariatric surgery (overall study) (Experimental): A prospective follow-up study is to estimate the prevalence of OSA and associated metabolic abnormalities in Finnish morbidly obese subjects and to evaluate the effects of bariatric surgery on OSA and associated metabolic abnormalities. The study is conducted in seven hospitals in Finland and 300 patients are planned to be recruited in the study.
  Interventions: Procedure: Bariatric surgery
- Bariatric surgery (randomised substudy) (Experimental): As a substudy of a larger trial, a randomized study on the effects of bariatric surgery compared to CPAP treatment will be performed in obese (BMI 35-45) patients with OSA. The included 100 (15/center) patients are randomised to two groups: surgical intervention group (50) and CPAP group (50). Patients in the surgical intervention group undergo standardised surgical treatment (laparoscopic gastric bypass), including general health information, such as avoidance of smoking, alcohol drinking, and importance of healthy nutrition and regular exercise. The CPAP group will be assigned to CPAP treatment and they also receive the general health information.
  Interventions: Procedure: Bariatric surgery
- CPAP (randomised substudy) (Active Comparator): As a substudy of a larger trial, a randomized study on the effects of bariatric surgery compared to CPAP treatment will be performed in obese (BMI 35-45) patients with OSA. The included 100 patients are randomised to two groups: surgical intervention group (50) and CPAP group (50). Patients in the surgical intervention group undergo standardised surgical treatment (laparoscopic gastric bypass), including general health information, such as avoidance of smoking, alcohol drinking, and importance of healthy nutrition and regular exercise. The CPAP group will be assigned to CPAP treatment and they also receive the general health information.
  Interventions: Device: Continuous positive airway pressure

INTERVENTIONS:
Procedure: Bariatric surgery — A standardized laparoscopic gastric bypass using Roux-en-Y technique
  Arms: Bariatric surgery (overall study); Bariatric surgery (randomised substudy)
Device: Continuous positive airway pressure — The patients are given standardized CPAP treatment according to current clinical guidelines.
  Arms: CPAP (randomised substudy)

SUMMARY:
Obesity is an increasing problem worldwide. Over 20% of people in western societies are obese (BMI >30kg/m2) and 1-2 % are morbidly obese (BMI >40 kg/m2). According to the recent study 6.6% of Finns are severely obese (BMI > 35kg/m2) and 2.0% are morbidly obese (BMI>40kg/m2). Because conventional treatments often fail to induce sustained weight loss obesity surgery has increased rapidly in many countries. Currently, > 300000 procedures are performed in the US each year. Thus in many European countries, including Finland, the need for obesity surgery is rapidly increasing.

The most important risk factor also for obstructive sleep apnea (OSA) is obesity, and thus effective treatment of obesity is the first-line treatment of OSA. However, Reliable information of the prevalence of OSA in morbidly obese patients is still lacking. The current knowledge is based on small studies, which have demonstrated that the prevalence of OSA may be higher than believed, even 70-80% in morbidly obese patients. There is a definite need for large, well-designed, prospective clinical studies to evaluate the effects of weight reduction in OSA and other co-morbidities related to obesity. Ever increasing research data showing a strong link between obesity and OSA and their co-existence as a major risk factor in the development of cardiovascular diseases should provoke concepts to search better clinical guidelines of diagnostics and treatments in a risk group, such as morbidly obese patients.

DETAILED DESCRIPTION:
Sleep disturbances have become a public health concern in the modern society, affecting millions of people. Obstructive sleep apnea (OSA) is one of the commonest sleep disturbances. Obstructive sleep apnea affects mostly middle-aged work force, causing a negative impact on public health since it increases both mortality and morbidity. In Finland, there are approximately 150,000 OSA patients, of whom 15,000 patients have a severe, 50,000 a moderate and 85,000 a mild form of the disease. The number of the patients is assumed to be strongly underestimated and it has been estimated that one out of five adults has at least mild OSA. OSA is tightly linked with metabolic abnormalities that contribute to an increased morbidity and mortality through cardiovascular disease. In addition, accidents by daytime sleepiness deteriorate person's quality of life and working capacity.

The most important risk factor for OSA is obesity, and thus effective treatment of obesity is first-line treatment of OSA. In a recent study it was observed that lifestyle intervention with an early weight reduction can be a curative treatment is mild OSA. However, regardless of these promising results weight reduction as a treatment of OSA is still underestimated. Particularly alarming is the exploding prevalence of morbid obesity, and that estimations have predicted this group of patients to increase most rapidly. Unfortunately, conventional lifestyle and weight reduction interventions have proven to be ineffective in long-term follow-up in these patients. In contrast, the permanent weight reduction achieved by bariatric surgery has been found to have favourable effects on diabetes, hyperlipidemia, hypertension, and also on OSA.

The treatment of OSA is demanding for both patients and physicians. There are no simple treatment modalities. Thus, there exists a definite need to improve the existing treatment modalities and to search new ones. The golden standard for treating patients with OSA is nasal continuous airway pressure (CPAP). It has been found to effective, but somewhat poor adherence (40-50%) to the treatment is certainly a major limitation. Moreover, there is little evidence about the possible beneficial metabolic effects of CPAP. Considering the rapid increase of obesity and the unsatisfactory adherence to CPAP treatment, bariatric surgery offers an interesting and viable option alongside with the conventional treatment modalities of OSA. Reliable information of the prevalence of OSA in morbidly obese patients is still lacking. The current knowledge is based on small studies, which have demonstrated that the prevalence of OSA could be higher than believed, even 70-80% in morbidly obese patients. There is a definite need for large, well-designed, prospective clinical studies on the effects of weight reduction in OSA and other co-morbidities related to obesity. Ever increasing research data showing a strong link between obesity and OSA and OSA as a major risk factor in the development of cardiovascular diseases should provoke concepts to improve better clinical guidelines of diagnostics and treatments in a risk group, such as obese patients.

ELIGIBILITY:
Inclusion Criteria:

For the overall study:

1. Age 18-65 years
2. BMI 35 and over with comorbidity (such as sleep apnea)
3. BMI 40 and over without any comorbidities
4. Obtained written consent

Additionally for the randomised substudy:

1. BMI 35-45
2. AHI 5-30

Exclusion Criteria:

1. On-going active treatment of OSA of any kind (during the last 1 month)
2. Pregnancy
3. Alcoholism
4. Eating disorders or severe depression
5. Other severe diseases contra-indicating bariatric surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The effect of bariatric surgery as a treatment of OSA | 1- and 5-year follow-up
  To evaluate the effect of bariatric surgery as a treatment of OSA measured by objective (cardio-respiratory recording) and subjective parameters (questionnaires).

SECONDARY OUTCOMES:
The prevalence of OSA in morbidly obese patients undergoing bariatric surgery | At the baseline
  To detect the prevalence of OSA in morbidly obese patients undergoing bariatric surgery in Finland.
The effect of bariatric surgery compared with CPAP treatment as a treatment of OSA | 6-month follow-up
  To evaluate the effect of bariatric surgery compared with CPAP treatment as a treatment of OSA measured by objective (cardio-respiratory recording) and subjective (questionnaires) parameters.
The effect of surgically induced weight loss on metabolism. | 3-, 6-, 12-, 60-month follow-up
  To study the effect of surgically induced weight loss on glucose tolerance, insulin resistance and lipid and energy metabolism.
The effect of weight loss on low-grade inflammation and peripheral blood mononuclear cells (PBMCs) gene expression | 3-, 6-, 12-, 60-month follow-up
  To study the effect of weight loss on OSA, low-grade inflammation and peripheral blood mononuclear cells (PBMCs) gene expression
The postoperative recovery after bariatric surgery | 3-, 6-, 12-, 60-month follow-up
  To evaluate the postoperative recovery after bariatric surgery
The effect of CPAP treatment on metabolism in morbidly obese patients with OSA | 3-, 6-month follow-up
  To evaluate the effect of CPAP treatment on metabolism in obese patients with OSA
The effect of CPAP treatment combined with bariatric surgery in obese patients with OSA. | 1- and 5-year follow-up
  To evaluate the effect of CPAP treatment combined with bariatric surgery in obese patients with OSA.

CONTACTS AND LOCATIONS:
Overall Officials: Henri Tuomilehto, MD, PhD, Study Director — Kuopio University Hospital; Mikael Victorzon, MD, PhD, Principal Investigator — Vaasa Central Hospital, Vaasa, Finland; Jussi Pihlajamäki, MD, PhD, Principal Investigator — Kuopio University Hospital
Locations (9):
- Finland (9):
  - Helsinki University hospital, Helsinki
  - National Institute for Health and Welfare, Helsinki
  - Helsinki Sleep Center, Helsinki
  - Eastern Finland Laboratory Centre, Kuopio
  - Kuopio University hospital, Kuopio
  - Päijät-Häme Central hospital, Lahti
  - Oulu University hospital, Oulu
  - Turku University hospital, Turku
  - Vaasa Central hospital, Vaasa

REFERENCES:
- [Derived] Peromaa-Haavisto P, Tuomilehto H, Kossi J, Virtanen J, Luostarinen M, Pihlajamaki J, Kakela P, Victorzon M. Obstructive sleep apnea: the effect of bariatric surgery after 12 months. A prospective multicenter trial. Sleep Med. 2017 Jul;35:85-90. doi: 10.1016/j.sleep.2016.12.017. Epub 2017 Jan 12. PMID 28549834